CLINICAL TRIAL: NCT01814410
Title: A Laboratory Study on the Interactive Effects of IV Ethanol and IV Nicotine on Subjective Effects and Cognition
Brief Title: Interactive Effects of IV Ethanol and IV Nicotine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: South Central VA Mental Illness Research, Education & Clinical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1209010841
Record Dates: First submitted 2013-01-18; First posted 2013-03-20 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Intravenous Ethanol; Intravenous Nicotine; Interactive effects; cognition; subjective effects; healthy subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- intravenous ethanol placebo and nicotine infusions (Placebo Comparator): Each subject will participate in three separate interventions. Each intervention will include three nicotine infusions (placebo and 2 active conditions). The interventions will differ on the ethanol infusion: placebo or one of two ethanol concentrations.
  Interventions: Drug: Intravenous ethanol placebo plus nicotine infusions
- intravenous ethanol 40% and nicotine infusions (Active Comparator): Each subject will participate in three separate interventions. Each intervention will include three nicotine infusions (placebo and 2 active conditions). The interventions will differ on the ethanol infusion: placebo or one of two ethanol concentrations.
  Interventions: Drug: intravenous ethanol 40mg% plus nicotine infusions
- intravenous ethanol 100% and nicotine infusions (Active Comparator): Each subject will participate in three separate interventions. Each intervention will include three nicotine infusions (placebo and 2 active conditions). The interventions will differ on the ethanol infusion: placebo or one of two ethanol concentrations.
  Interventions: Drug: intravenous ethanol 100mg% plus nicotine infusions

INTERVENTIONS:
Drug: Intravenous ethanol placebo plus nicotine infusions — nicotine infusions: 1) placebo; 2) nicotine 0.5 mg/70 kg; 3) nicotine 1.0 mg/70 kg
  Arms: intravenous ethanol placebo and nicotine infusions
Drug: intravenous ethanol 40mg% plus nicotine infusions — nicotine infusions: 1) placebo; 2) nicotine 0.5 mg/70 kg; 3) nicotine 1.0 mg/70 kg
  Arms: intravenous ethanol 40% and nicotine infusions
Drug: intravenous ethanol 100mg% plus nicotine infusions — nicotine infusions: 1) placebo; 2) nicotine 0.5 mg/70 kg; 3) nicotine 1.0 mg/70 kg
  Arms: intravenous ethanol 100% and nicotine infusions

SUMMARY:
There are mixed reports on nicotine's effects on ethanol-induced impairment in cognitive performance and behavior in humans. The main objective of this study is to characterize the interactive effects of acute intravenous (IV) ethanol and nicotine administration on cognition and behavior in healthy smokers. The general hypothesis is that nicotine will attenuate the negative effects of ethanol on cognition and subjective stimulant/sedative effects of ethanol.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female;
2. between the ages of 21 and 50 years;
3. medically and neurologically healthy on the basis of history, physical examination, EKG, screening laboratories
4. history of smoking daily for the past 12 months, at least 5 cigarettes daily; not seeking treatment for nicotine dependence
5. social drinkers no maximum level of alcohol consumption will be defined a priori but individuals who met current DSM -IV criteria for alcohol dependence (abuse will be allowed) will be excluded from the study.

Exclusion Criteria:

1. history of major medical illnesses that the physician investigator deems as contraindicated for the patient to be in the study;
2. regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and recent psychiatric diagnosis and treatment for Axis I disorders including major depression, bipolar affective disorder, schizophrenia or panic disorder;
3. current abuse of any recreational or prescription drugs (except alcohol);
4. alcohol naïve.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Biphasic Alcohol Effects Scale (BAES) | 2 minutes
  A 14-item scale with 7 items designed to assess stimulant effects associated with the ascending limb of ethanol intoxication and 7 items developed to measure sedative effects associated with the descending limb of ethanol intoxication.

SECONDARY OUTCOMES:
Visual Analog Scales of Mood States | 1 minute
  The following items will be assessed: high, depressed, anxious, drowsy, irritable, tired, sad, angry, nervous, nauseous, blurred vision, flushed, headache, lightheaded, dizzy, sweating, abdominal discomfort and tingling .
QSU-Brief | 2 minutes
  A measure of smoking urges reflecting not only intent and desire to smoke, and anticipation of pleasure from smoking, but also anticipation of relief from negative affect and nicotine withdrawal, and urgent and overwhelming desire to smoke.
Digit Symbol Substitution Task | 2 minutes
  A test of psychomotor performance, which measures motor persistence, sustained attention, response speed and visuomotor coordination.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ralevski, Ph.D., Principal Investigator — Yale University
Locations (1):
- West Haven VA Hospital, West Haven, Connecticut, United States